CLINICAL TRIAL: NCT03538899
Title: A Phase I/II Safety and Efficacy Study of Gene Transfer for Artemis-Deficient Severe Combined Immunodeficiency (ART-SCID) in Newly Diagnosed Patients Using a Self-Inactivating Lentiviral Vector (AProArt) to Transduce Autologous CD34 Hematopoietic Cells (AProArt-CD34)
Brief Title: Autologous Gene Therapy for Artemis-Deficient SCID
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Morton Cowan, Professor Emeritus, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-22799; CLIN2-10830 (Other Grant/Funding Number: California Institute of Regenerative Medicine); CLIN2-17127 (Other Grant/Funding Number: California Institute of Regenerative Medicine)
Record Dates: First submitted 2018-05-03; First posted 2018-05-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Artemis-deficient Severe Combined Immunodeficiency; gene therapy; autologous stem cell transplant
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Busulfan

STUDY DESIGN:
Intervention Model Description: Longitudinal study of autologous stem cell transplant of cells transduced with corrected DCLRE1C gene using a self-inactivating lentiviral vector (AProArt). The CliniMACS® CD34 Reagent System cell sorter device will be used to select CD 34 cells. Sub-ablative busulfan will be used for pre-transplant conditioning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Gene therapy (AProArt) (Experimental): Gene Transfer for Artemis-Deficient Severe Combined Immunodeficiency (ART-SCID) Using a Self-Inactivating Lentiviral Vector (AProArt) to Transduce Autologous CD34 Hematopoietic Cells. The CliniMACS® CD34 Reagent System sorter device will be used to select CD34 cells. Patients will be conditioned with low dose busulfan prior to transplant.
  Interventions: Drug: AProArt-CD34; Device: CliniMACS® CD34 Reagent System cell sorter device; Drug: Busulfan

INTERVENTIONS:
Drug: AProArt-CD34 — Participants will undergo infusion with autologous hematopoietic cells transduced with a lentiviral vector, AProArt, which contains the correct form of DCLRE1C complementary deoxyribonucleic acid DNA, after receiving sub-ablative, exposure-targeted busulfan conditioning.
  Other Names: lentiviral gene therapy using AProArt
Device: CliniMACS® CD34 Reagent System cell sorter device — Processing of hematopoietic progenitor cells to select CD34 cells, using the CliniMACS® CD34 Reagent System, prior to infusion.
Drug: Busulfan — Busulfan is a cell cycle non-specific alkylating antineoplastic agent, in the class of alkyl sulfonates. Patients will receive low-dose busulfan conditioning targeted over 2 days to achieve a cumulative area under the curve (AUC) of 20 mg*hr/L.
  Other Names: Busulfex

SUMMARY:
This study aims to determine if a new method can be used to treat Artemis-deficient Severe Combined Immunodeficiency (ART-SCID), a severe form of primary immunodeficiency caused by mutations in the DCLRE1C gene. This method involves transferring a normal copy of the DCLRE1C gene into stem cells of an affected patient. Participants will receive an infusion of stem cells transduced with a self-inactivating lentiviral vector that contains a normal copy of the DCLRE1C gene. Prior to the infusion they will receive sub-ablative, dose-targeted busulfan conditioning. The study will investigate if the procedure is safe, whether it can be done according to the methods described in the protocol, and whether the procedure will provide a normal immune system for the patient. A total of 24 newly diagnosed patients will be enrolled at the University of California San Francisco in this single-site trial and will be followed for 15 years post-infusion. It is hoped that this type of gene transfer may offer improved outcomes for ART-SCID patients who lack a brother or sister who can be used as a donor for stem cell transplantation or who have failed to develop a functioning immune system after a previous stem cell transplant.

DETAILED DESCRIPTION:
Children with SCID generally do not survive beyond the first year of life without definitive treatment. The most effective current cure is hematopoietic stem cell transplant (HCT) with a human leukocyte antigen (HLA) matched sibling. While a matched sibling HCT can successfully treat ART-SCID, fewer than 20% of affected children have such a donor, and even when a matched sibling donor is available there is often incomplete T and B cell immune reconstitution. ART-SCID is the most difficult type of SCID to cure by hematopoietic stem cell transplant using alternative donors. Engraftment typically requires intensive conditioning with high dose alkylating agents to prevent rejection and to open marrow niches. These patients also have a high risk of developing graft versus host disease (GVHD) when alternative donors are used. The great majority of patients have absent B cell reconstitution and require lifelong administration of immunoglobulin infusions. Patients with ART-SCID who do receive high doses of alkylators, especially when 2 agents are used, have poorer survival, abnormal dental development, endocrinopathies, and short stature in comparison with children exposed to no or limited alkylators or children with SCID types that are not associated with a DNA repair defect. For these reasons, a safer, more effective approach to curing ART-SCID is needed. Autologous gene-corrected hematopoeitic stem cell transplant may eliminate both the risk of GVHD and the need for alkylators to prevent rejection.

The study design is a single-cohort, longitudinal experiment using non-randomized patients treated once with a lentiviral vector for gene-correction of Artemis-deficient SCID after conditioning with low-dose busulfan. No formal control group is planned for gauging safety; rather, intensive monitoring of the initial 6 enrollees was undertaken to preclude continued accrual in the presence of safety signals. This enrollment stage was completed in 2019 with no safety signals identified, and long-term safety will be monitored for 15 years. Bone marrow stem cells will be harvested from participants, and CD34 cells will be isolated using the CliniMACS® CD34 Reagent System cell sorter device. The CD34 cells will be transduced with the AProArt lentiviral vector, and cryopreserved. Aliquots of the cells will undergo safety testing and be reserved for potency evaluation. All patients will receive busulfan conditioning targeted over 2 days to achieve a cumulative area under the curve (AUC) of 20 mg*hr/L (an ablative cumulative AUC is 60-90mg*hr/L).

Following the infusion of AProArt-transduced cells, patients will be assessed weekly through 12 weeks post-transplant and at week 16, monthly through month 6 post-transplant, every 3 months through month 24, every 6 months during years 2-5, and then annually through year 15. Assessments will include physical examination, clinical laboratory tests, collection of specimens for research studies, and completion of Quality of Life questionnaires. Neurodevelopmental testing will be performed at age-appropriate time points.

At weeks 4, 6, 8, 12, 16, and 24, research specimens will be evaluated for evidence of gene transduced peripheral blood mononuclear cells and when possible, cell lineages including T, B, NK and granulocyte/myeloid cells. If there is no evidence of gene transduced cells at 6 weeks (42 days) post infusion, planning for an alternative treatment will begin, with the final decision regarding further therapy to be based on gene-marking results at 10 weeks.

If the absolute neutrophil count is < 200/µl or platelets < 20,000/µl on 3 independent determinations after day 42 post infusion of transduced cells, the patient may receive an allogeneic hematopoeitic stem cell transplant. Patients who were neutropenic prior to conditioning (SCID-related neutropenia) but responsive to granulocyte-colony stimulating factor (GCSF) will not be considered to have failed, provided the absolute neutrophil count can be maintained above >300/µl with GCSF.

Recipients will be followed for toxicity and durable reconstitution of T and B cell immunity. Immune reconstitution of T cells will be monitored on a regular basis. Patients with evidence of clinically inadequate immune reconstitution, low vector copy number (VCN), or any other features suggesting clinically inadequate response to the initial gene therapy procedure will be offered a repeat infusion of gene-transduced cells. Conditioning regimens given prior to a repeat gene therapy procedure may include low-dose busulfan, other conditioning, or no conditioning.

Historical controls who received alternative donor allogeneic transplants as treatment for ART-SCID will serve as the comparator arm for secondary endpoints.

An independent Data Safety Monitoring Board (DSMB) has been appointed for safety monitoring of this trial. The DSMB reviews all data for safety on a regular schedule, based on numbers of enrolled subjects and conducts special urgent review of any protocol related Serious Adverse Events (SAE). In the early stage of the trial, the DSMB reviewed results of each of the first 3 cases prior to proceeding with subsequent patients.

The investigational product (IND17711) for the ART-SCID gene transfer study is not available for expanded access use. As per 21 CFR Part 312.305(3), the study management team has determined that providing the investigational product for expanded access use at this time would interfere with the conduct and completion of the clinical trial and potential development of future expanded access use. The investigational product is available to eligible patients through participation in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥2.0 months of age at initiation of busulfan conditioning
* New diagnosis of typical or minimally leaky ART-SCID, as defined by the criteria below:
* Artemis deficiency with bi-allelic pathogenic or likely pathogenic mutations in DCLRE1C; AND
* CD3 count < 50 autologous cells/µL (typical ART-SCID) OR spontaneous maternal chimerism, OR CD3 count >50/µL and <300/uL and with restricted T cell receptor Vb diversity; AND
* CD45 cell response to mitogens (PHA) < 50% of the lower limit of normal range for the lab (leaky ART-SCID).
* No medically eligible HLA-identical sibling with a normal immune system who could serve as an allogeneic bone marrow donor (applies to newly diagnosed patients only).

Exclusion Criteria:

* Presence of a medically eligible HLA-matched sibling
* Evidence of HIV infection by polymerase chain reaction or p24 antigen testing.
* Unable to tolerate general anesthesia and/or marrow harvest or insertion of central venous catheter.
* Any one of liver function tests AST, ALT, gamma-glutamyl transpeptidase (GGT) >5X the upper limit of normal for lab and/or total bilirubin >2.0 mg/dl (not due to Gilbert's) at the time of planned initiation of busulfan conditioning unless the elevated LFTs are considered to be due to medication, a viral infection for which there is no treatment other than reconstituting T cell immunity, or maternal GVHD.
* Presence of any severe medical conditions making a patient unsuitable for busulfan administration
* Presence of a recognized second gene mutation that results in an autosomal dominant or recessive disorder intrinsic to hematopoietic cells and that could be treated by an allogeneic HCT.
* Presence of a medical condition indicating that survival is predicted to be less than 4 months, such as the requirement for mechanical ventilation, severe failure of a major organ system, or evidence of a serious, progressive infection that is refractory to medical therapy.
* A social situation indicating that the family may not be able to comply with protocol procedures and recommended medical care and follow-up.
* Other conditions which in the opinion of the Principal Investigator and/or co-investigators, contra-indicate the infusion of transduced cells or study participation.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2038-06 (Estimated); Study Completion 2038-06 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that ART-SCID patients receiving AProArt-CD34 infusion have superior overall survival (OS) at 24 months post treatment with AProArt-CD34 versus the established outcome of 0% OS for patients who receive no treatment for ART-SCID | 24 months
  Patient survival status and (if applicable) cause of death will be recorded to assess overall survival.

SECONDARY OUTCOMES:
B cell immune reconstitution by 24±2 months compared with historical control cohort of allogeneic transplant recipients | 24 months
  B cell immune reconstitution will be defined as cessation of immunoglobulin replacement therapy
Number of participants with T cell immune reconstitution compared with historical controls who received allogeneic transplants to treat ART-SCID. | 24 months
  T cell immune reconstitution will be defined as presence of both of the following: 1) a. CD3>1000/mm3; 2) CD4>500/mm3.
Event Free Survival | 24 months
  Events are defined as death, use of a repeat infusion of gene-corrected cells to enhance T/B cell immune reconstitution or requirement for performance of an allogeneic HCT.

OTHER OUTCOMES:
Adverse event (AE) profile associated with the study intervention from treatment through 15 years after the gene transfer procedure | 15 years
  Clinical and laboratory AEs as measured by CTCAE V4
Number of participants with B cell reconstitution beyond 24 months, including B cell numbers and function | 15 years
  B cell reconstitution will be defined as presence of at least two of the following: 1) B cell number >40/mm3; 2) Cessation of immunoglobulin replacement therapy; 3) Protective specific antibody responses. The number of participants who meet the definition for B cell reconstitution will be tabulated.
Efficacy of targeting low exposure busulfan in infants and children, calculated by percentage of participants whose treatment meets study parameters using a validated population pharmacokinetic model to calculate individualized busulfan clearance. | 42 days
  Achievement of final target cumulative AUC of 20±2 mg*hr/L in approximately 90% of subjects
Repertoire diversity of T and B cells, as assessed by analyzing T cell receptor gene variable beta sequence (TCR-Vb) and immunoglobulin heavy chain (IGH) rearranged receptors and calculating diversity Shannon Index. | 24 months
  Measured by deep sequencing of the T cell receptor (TCR) gene variable beta sequence (TCR-Vb) and immunoglobulin heavy chain (IGH) rearranged receptors. The diversity Shannon Index is expected to be above 7.5 by 24±2 months post treatment in 90% of patients.
Determine if B cell receptor diversity at 6 months is predictive of B cell reconstitution over 15 years by analyzing B cell receptor gene variable beta sequence and immunoglobulin heavy chain rearranged receptors and calculating diversity Shannon Index. | 15 years
  A Shannon Index >5 is expected to be a biomarker for B cell reconstitution. B cell receptor diversity will be measured throughout study participation.
Determine if at 6 months T cell receptor (TCR) diversity and/or absolute CD3, CD4, naïve CD4 counts predict T cell reconstitution at 24 months or need for 2nd treatment throughout the 15 year follow-up period. | 15 years
  TCR-Vb diversity and absolute CD3, CD4 and naïve CD4 counts will be measured at 6 months. T cell reconstitution will be measured throughout study participation.
Stability of mean vector copy number (VCN) and the location of vector integration sites in sorted T, B, and natural killer (NK) cells, granulocytes and monocytes in peripheral blood over time after infusion of transduced HSC. | 24 months
  Mean vector copy number (VCN) and the location of vector integration sites will be measured at 6±1, 12±1 and 24±2 months and then annually through 15 years after infusion of AProArt-CD34. The mean VCN should be >0.5 copies/cell in T and B cells and >0.01 in NK, myeloid and granulocytes by 24±2 months post treatment.
Characterization of insertion sites in multiple cell lineages as an indicator of diversity, multilineage engraftment, and tabulation of any clonal expansion that might indicate development of a malignancy. | 24 months
  Insertion sites will be measured at 6±1, 12±1, 24±2 months, and annually through 15 years after infusion of AProArt-CD34. Cell insertion sites are expected to be diverse with no clone representing >20% of a lineage at 24 months.
Potential benefit of prophylactic sirolimus in reducing the incidence of transient autoimmune hemolytic anemia (AIHA) post infusion of AProArt-CD34, as assessed by number of participants with clinical diagnosis of AIHA. | 24 months
  Incidence of autoimmune hemolytic anemia by 24±2 months post infusion following administration of prophylactic sirolimus, as assessed by monitoring of hemoglobin, direct and indirect Coombs, reticulocyte, and lactate dehydrogenase results. Incidence of AIHA requiring treatment is expected to be <40% of patients on prophylactic sirolimus.
Measurement of radiation sensitivity in peripheral blood NK cells for development and validation of a rapid functional assay for radiation-sensitive SCID. | 24 months
  Development and validation of an assay for radiation sensitive SCID in peripheral blood NK cells
Potency of AProArt-CD34 as indicated by capacity for in vitro differentiation of participant specimens into T cells and assessment of average VCN as a surrogate marker for potency. | 5 years
  Demonstration that post-transduction patient CD34+ cells have the capacity for in vitro differentiation into T cells and that average VCN is a surrogate marker for potency. One or more potency assays will be developed and validated for AProArt-transduced CD34+ HSC that give results within 52 days of transduction, and correlation of these with VCN obtained at 6 and 14 days post transduction with AProArt.
Hematopoietic recovery in patients with ART-SCID who receive self-inactivating (SIN) lentiviral vector (AProArt)-transduced CD34 cells through a repeat infusion autologous stem cell transplant. | 5 years
  Patients will undergo blood tests to measure complete blood count and differential following a repeat infusion of gene corrected cells.
Effects of targeted low exposure busulfan conditioning on patient growth/stature | 5 years
  Patient growth will be compared with norms for age
Effects of busulfan on patient dental development | 5 years
  Dental development will be compared with normal development of permanent teeth from age 5 through age 15 years
Patient reported outcome of undergoing treatment with gene-corrected cells as assessed by the PedsQL questionnaires. | 5 years
  Age-appropriate PedsQL questionnaires will be administered at baseline and years 1, 2, 4, 8, 10, 12, and 15.
Family impact of undergoing treatment with gene-corrected cells. | 15 years
  The PedsQL Family Impact module will be administered at baseline and years 1, 2, 4, 8, 10, 12, and 15.
Effects of the study intervention on neurodevelopment over time | 5 years
  Neurodevelopment test results will be compared with norms for ages 18 months and ages 3, 5, 8, 11, 14 and 17 years.

CONTACTS AND LOCATIONS:
Overall Officials: Morton Cowan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco (UCSF) Children's Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in scientific journals (text, tables, figures, and appendices) after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers can submit a request for access to the study Steering Committee. If the proposal is determined to be methodologically sound, data requestors will need to sign a data access agreement prior to gaining access.

REFERENCES:
- [Background] Buckley RH. The multiple causes of human SCID. J Clin Invest. 2004 Nov;114(10):1409-11. doi: 10.1172/JCI23571. PMID 15545990
- [Background] Gatti RA, Meuwissen HJ, Allen HD, Hong R, Good RA. Immunological reconstitution of sex-linked lymphopenic immunological deficiency. Lancet. 1968 Dec 28;2(7583):1366-9. doi: 10.1016/s0140-6736(68)92673-1. No abstract available. PMID 4177932
- [Background] Chan A, Scalchunes C, Boyle M, Puck JM. Early vs. delayed diagnosis of severe combined immunodeficiency: a family perspective survey. Clin Immunol. 2011 Jan;138(1):3-8. doi: 10.1016/j.clim.2010.09.010. Epub 2010 Oct 28. PMID 21035402
- [Background] Chan K, Puck JM. Development of population-based newborn screening for severe combined immunodeficiency. J Allergy Clin Immunol. 2005 Feb;115(2):391-8. doi: 10.1016/j.jaci.2004.10.012. PMID 15696101
- [Background] Kwan A, Puck JM. History and current status of newborn screening for severe combined immunodeficiency. Semin Perinatol. 2015 Apr;39(3):194-205. doi: 10.1053/j.semperi.2015.03.004. Epub 2015 Apr 30. PMID 25937517
- [Background] Pai SY, Logan BR, Griffith LM, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Hanson IC, Filipovich AH, Jyonouchi S, Sullivan KE, Small TN, Burroughs L, Skoda-Smith S, Haight AE, Grizzle A, Pulsipher MA, Chan KW, Fuleihan RL, Haddad E, Loechelt B, Aquino VM, Gillio A, Davis J, Knutsen A, Smith AR, Moore TB, Schroeder ML, Goldman FD, Connelly JA, Porteus MH, Xiang Q, Shearer WT, Fleisher TA, Kohn DB, Puck JM, Notarangelo LD, Cowan MJ, O'Reilly RJ. Transplantation outcomes for severe combined immunodeficiency, 2000-2009. N Engl J Med. 2014 Jul 31;371(5):434-46. doi: 10.1056/NEJMoa1401177. PMID 25075835
- [Background] Dorsey MJ, Dvorak CC, Cowan MJ, Puck JM. Treatment of infants identified as having severe combined immunodeficiency by means of newborn screening. J Allergy Clin Immunol. 2017 Mar;139(3):733-742. doi: 10.1016/j.jaci.2017.01.005. PMID 28270365
- [Background] Dvorak CC, Hassan A, Slatter MA, Honig M, Lankester AC, Buckley RH, Pulsipher MA, Davis JH, Gungor T, Gabriel M, Bleesing JH, Bunin N, Sedlacek P, Connelly JA, Crawford DF, Notarangelo LD, Pai SY, Hassid J, Veys P, Gennery AR, Cowan MJ. Comparison of outcomes of hematopoietic stem cell transplantation without chemotherapy conditioning by using matched sibling and unrelated donors for treatment of severe combined immunodeficiency. J Allergy Clin Immunol. 2014 Oct;134(4):935-943.e15. doi: 10.1016/j.jaci.2014.06.021. Epub 2014 Aug 7. PMID 25109802
- [Background] Neven B, Leroy S, Decaluwe H, Le Deist F, Picard C, Moshous D, Mahlaoui N, Debre M, Casanova JL, Dal Cortivo L, Madec Y, Hacein-Bey-Abina S, de Saint Basile G, de Villartay JP, Blanche S, Cavazzana-Calvo M, Fischer A. Long-term outcome after hematopoietic stem cell transplantation of a single-center cohort of 90 patients with severe combined immunodeficiency. Blood. 2009 Apr 23;113(17):4114-24. doi: 10.1182/blood-2008-09-177923. Epub 2009 Jan 23. PMID 19168787
- [Background] Schuetz C, Neven B, Dvorak CC, Leroy S, Ege MJ, Pannicke U, Schwarz K, Schulz AS, Hoenig M, Sparber-Sauer M, Gatz SA, Denzer C, Blanche S, Moshous D, Picard C, Horn BN, de Villartay JP, Cavazzana M, Debatin KM, Friedrich W, Fischer A, Cowan MJ. SCID patients with ARTEMIS vs RAG deficiencies following HCT: increased risk of late toxicity in ARTEMIS-deficient SCID. Blood. 2014 Jan 9;123(2):281-9. doi: 10.1182/blood-2013-01-476432. Epub 2013 Oct 21. PMID 24144642
- [Background] Wahlstrom JT, Dvorak CC, Cowan MJ. Hematopoietic Stem Cell Transplantation for Severe Combined Immunodeficiency. Curr Pediatr Rep. 2015 Mar 1;3(1):1-10. doi: 10.1007/s40124-014-0071-7. PMID 25821657
- [Background] Horn B, Cowan MJ. Unresolved issues in hematopoietic stem cell transplantation for severe combined immunodeficiency: need for safer conditioning and reduced late effects. J Allergy Clin Immunol. 2013 May;131(5):1306-11. doi: 10.1016/j.jaci.2013.03.014. PMID 23622119
- [Background] Cowan MJ, Gennery AR. Radiation-sensitive severe combined immunodeficiency: The arguments for and against conditioning before hematopoietic cell transplantation--what to do? J Allergy Clin Immunol. 2015 Nov;136(5):1178-85. doi: 10.1016/j.jaci.2015.04.027. Epub 2015 Jun 6. PMID 26055221
- [Background] Cicalese MP, Aiuti A. Clinical applications of gene therapy for primary immunodeficiencies. Hum Gene Ther. 2015 Apr;26(4):210-9. doi: 10.1089/hum.2015.047. PMID 25860576
- [Background] Cavazzana-Calvo M, Fischer A. Gene therapy for severe combined immunodeficiency: are we there yet? J Clin Invest. 2007 Jun;117(6):1456-65. doi: 10.1172/JCI30953. PMID 17549248
- [Background] Hacein-Bey-Abina S, Pai SY, Gaspar HB, Armant M, Berry CC, Blanche S, Bleesing J, Blondeau J, de Boer H, Buckland KF, Caccavelli L, Cros G, De Oliveira S, Fernandez KS, Guo D, Harris CE, Hopkins G, Lehmann LE, Lim A, London WB, van der Loo JC, Malani N, Male F, Malik P, Marinovic MA, McNicol AM, Moshous D, Neven B, Oleastro M, Picard C, Ritz J, Rivat C, Schambach A, Shaw KL, Sherman EA, Silberstein LE, Six E, Touzot F, Tsytsykova A, Xu-Bayford J, Baum C, Bushman FD, Fischer A, Kohn DB, Filipovich AH, Notarangelo LD, Cavazzana M, Williams DA, Thrasher AJ. A modified gamma-retrovirus vector for X-linked severe combined immunodeficiency. N Engl J Med. 2014 Oct 9;371(15):1407-17. doi: 10.1056/NEJMoa1404588. PMID 25295500
- [Background] Greene MR, Lockey T, Mehta PK, Kim YS, Eldridge PW, Gray JT, Sorrentino BP. Transduction of human CD34+ repopulating cells with a self-inactivating lentiviral vector for SCID-X1 produced at clinical scale by a stable cell line. Hum Gene Ther Methods. 2012 Oct;23(5):297-308. doi: 10.1089/hgtb.2012.150. Epub 2012 Nov 7. PMID 23075105
- [Background] De Ravin SS, Wu X, Moir S, Anaya-O'Brien S, Kwatemaa N, Littel P, Theobald N, Choi U, Su L, Marquesen M, Hilligoss D, Lee J, Buckner CM, Zarember KA, O'Connor G, McVicar D, Kuhns D, Throm RE, Zhou S, Notarangelo LD, Hanson IC, Cowan MJ, Kang E, Hadigan C, Meagher M, Gray JT, Sorrentino BP, Malech HL, Kardava L. Lentiviral hematopoietic stem cell gene therapy for X-linked severe combined immunodeficiency. Sci Transl Med. 2016 Apr 20;8(335):335ra57. doi: 10.1126/scitranslmed.aad8856. PMID 27099176
- [Background] Kwan A, Hu D, Song M, Gomes H, Brown DR, Bourque T, Gonzalez-Espinosa D, Lin Z, Cowan MJ, Puck JM. Successful newborn screening for SCID in the Navajo Nation. Clin Immunol. 2015 May;158(1):29-34. doi: 10.1016/j.clim.2015.02.015. Epub 2015 Mar 8. PMID 25762520
- [Background] Li L, Drayna D, Hu D, Hayward A, Gahagan S, Pabst H, Cowan MJ. The gene for severe combined immunodeficiency disease in Athabascan-speaking Native Americans is located on chromosome 10p. Am J Hum Genet. 1998 Jan;62(1):136-44. doi: 10.1086/301688. PMID 9443881
- [Background] Li L, Moshous D, Zhou Y, Wang J, Xie G, Salido E, Hu D, de Villartay JP, Cowan MJ. A founder mutation in Artemis, an SNM1-like protein, causes SCID in Athabascan-speaking Native Americans. J Immunol. 2002 Jun 15;168(12):6323-9. doi: 10.4049/jimmunol.168.12.6323. PMID 12055248
- [Background] Li L, Salido E, Zhou Y, Bhattacharyya S, Yannone SM, Dunn E, Meneses J, Feeney AJ, Cowan MJ. Targeted disruption of the Artemis murine counterpart results in SCID and defective V(D)J recombination that is partially corrected with bone marrow transplantation. J Immunol. 2005 Feb 15;174(4):2420-8. doi: 10.4049/jimmunol.174.4.2420. PMID 15699179
- [Background] Xiao Z, Dunn E, Singh K, Khan IS, Yannone SM, Cowan MJ. A non-leaky Artemis-deficient mouse that accurately models the human severe combined immune deficiency phenotype, including resistance to hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2009 Jan;15(1):1-11. doi: 10.1016/j.bbmt.2008.10.026. PMID 19135937
- [Background] Multhaup M, Karlen AD, Swanson DL, Wilber A, Somia NV, Cowan MJ, McIvor RS. Cytotoxicity associated with artemis overexpression after lentiviral vector-mediated gene transfer. Hum Gene Ther. 2010 Jul;21(7):865-75. doi: 10.1089/hum.2009.162. PMID 20163250
- [Background] Multhaup MM, Podetz-Pedersen KM, Karlen AD, Olson ER, Gunther R, Somia NV, Blazar BR, Cowan MJ, McIvor RS. Role of transgene regulation in ex vivo lentiviral correction of artemis deficiency. Hum Gene Ther. 2015 Apr;26(4):232-43. doi: 10.1089/hum.2014.062. Epub 2015 Apr 13. PMID 25738323
- [Background] Punwani D, Kawahara M, Yu J, Sanford U, Roy S, Patel K, Carbonaro DA, Karlen AD, Khan S, Cornetta K, Rothe M, Schambach A, Kohn DB, Malech HL, McIvor RS, Puck JM, Cowan MJ. Lentivirus Mediated Correction of Artemis-Deficient Severe Combined Immunodeficiency. Hum Gene Ther. 2017 Jan;28(1):112-124. doi: 10.1089/hum.2016.064. Epub 2016 Sep 7. PMID 27611239
- [Background] Yeager AM, Shinn C, Shinohara M, Pardoll DM. Hematopoietic cell transplantation in the twitcher mouse. The effects of pretransplant conditioning with graded doses of busulfan. Transplantation. 1993 Jul;56(1):185-90. doi: 10.1097/00007890-199307000-00034. PMID 8101401
- [Background] Modlich U, Navarro S, Zychlinski D, Maetzig T, Knoess S, Brugman MH, Schambach A, Charrier S, Galy A, Thrasher AJ, Bueren J, Baum C. Insertional transformation of hematopoietic cells by self-inactivating lentiviral and gammaretroviral vectors. Mol Ther. 2009 Nov;17(11):1919-28. doi: 10.1038/mt.2009.179. Epub 2009 Aug 11. PMID 19672245
- [Background] O'Marcaigh AS, DeSantes K, Hu D, Pabst H, Horn B, Li L, Cowan MJ. Bone marrow transplantation for T-B- severe combined immunodeficiency disease in Athabascan-speaking native Americans. Bone Marrow Transplant. 2001 Apr;27(7):703-9. doi: 10.1038/sj.bmt.1702831. PMID 11360109
- [Background] Grunebaum E, Roifman CM. Bone marrow transplantation using HLA-matched unrelated donors for patients suffering from severe combined immunodeficiency. Immunol Allergy Clin North Am. 2010 Feb;30(1):63-73. doi: 10.1016/j.iac.2009.11.001. PMID 20113887
- [Background] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Pai SY, Ballard B, Bauer SC, Bleesing JJ, Boyle M, Brower A, Buckley RH, van der Burg M, Burroughs LM, Candotti F, Cant AJ, Chatila T, Cunningham-Rundles C, Dinauer MC, Dvorak CC, Filipovich AH, Fleisher TA, Bobby Gaspar H, Gungor T, Haddad E, Hovermale E, Huang F, Hurley A, Hurley M, Iyengar S, Kang EM, Logan BR, Long-Boyle JR, Malech HL, McGhee SA, Modell F, Modell V, Ochs HD, O'Reilly RJ, Parkman R, Rawlings DJ, Routes JM, Shearer WT, Small TN, Smith H, Sullivan KE, Szabolcs P, Thrasher A, Torgerson TR, Veys P, Weinberg K, Zuniga-Pflucker JC; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) report. J Allergy Clin Immunol. 2014 Feb;133(2):335-47. doi: 10.1016/j.jaci.2013.07.052. Epub 2013 Oct 15. PMID 24139498
- [Background] Ferrua F, Brigida I, Aiuti A. Update on gene therapy for adenosine deaminase-deficient severe combined immunodeficiency. Curr Opin Allergy Clin Immunol. 2010 Dec;10(6):551-6. doi: 10.1097/ACI.0b013e32833fea85. PMID 20966749
- [Background] Candotti F, Shaw KL, Muul L, Carbonaro D, Sokolic R, Choi C, Schurman SH, Garabedian E, Kesserwan C, Jagadeesh GJ, Fu PY, Gschweng E, Cooper A, Tisdale JF, Weinberg KI, Crooks GM, Kapoor N, Shah A, Abdel-Azim H, Yu XJ, Smogorzewska M, Wayne AS, Rosenblatt HM, Davis CM, Hanson C, Rishi RG, Wang X, Gjertson D, Yang OO, Balamurugan A, Bauer G, Ireland JA, Engel BC, Podsakoff GM, Hershfield MS, Blaese RM, Parkman R, Kohn DB. Gene therapy for adenosine deaminase-deficient severe combined immune deficiency: clinical comparison of retroviral vectors and treatment plans. Blood. 2012 Nov 1;120(18):3635-46. doi: 10.1182/blood-2012-02-400937. Epub 2012 Sep 11. PMID 22968453
- [Background] Multhaup MM, Gurram S, Podetz-Pedersen KM, Karlen AD, Swanson DL, Somia NV, Hackett PB, Cowan MJ, McIvor RS. Characterization of the human artemis promoter by heterologous gene expression in vitro and in vivo. DNA Cell Biol. 2011 Oct;30(10):751-61. doi: 10.1089/dna.2011.1244. Epub 2011 Jun 10. PMID 21663454
- [Background] Heimall J, Puck J, Buckley R, Fleisher TA, Gennery AR, Neven B, Slatter M, Haddad E, Notarangelo LD, Baker KS, Dietz AC, Duncan C, Pulsipher MA, Cowan MJ. Current Knowledge and Priorities for Future Research in Late Effects after Hematopoietic Stem Cell Transplantation (HCT) for Severe Combined Immunodeficiency Patients: A Consensus Statement from the Second Pediatric Blood and Marrow Transplant Consortium International Conference on Late Effects after Pediatric HCT. Biol Blood Marrow Transplant. 2017 Mar;23(3):379-387. doi: 10.1016/j.bbmt.2016.12.619. Epub 2017 Jan 6. PMID 28068510
- [Background] Pai SY, Cowan MJ. Stem cell transplantation for primary immunodeficiency diseases: the North American experience. Curr Opin Allergy Clin Immunol. 2014 Dec;14(6):521-6. doi: 10.1097/ACI.0000000000000115. PMID 25259542
- [Background] Hacein-Bey-Abina S, Hauer J, Lim A, Picard C, Wang GP, Berry CC, Martinache C, Rieux-Laucat F, Latour S, Belohradsky BH, Leiva L, Sorensen R, Debre M, Casanova JL, Blanche S, Durandy A, Bushman FD, Fischer A, Cavazzana-Calvo M. Efficacy of gene therapy for X-linked severe combined immunodeficiency. N Engl J Med. 2010 Jul 22;363(4):355-64. doi: 10.1056/NEJMoa1000164. PMID 20660403
- [Background] Hacein-Bey Abina S, Gaspar HB, Blondeau J, Caccavelli L, Charrier S, Buckland K, Picard C, Six E, Himoudi N, Gilmour K, McNicol AM, Hara H, Xu-Bayford J, Rivat C, Touzot F, Mavilio F, Lim A, Treluyer JM, Heritier S, Lefrere F, Magalon J, Pengue-Koyi I, Honnet G, Blanche S, Sherman EA, Male F, Berry C, Malani N, Bushman FD, Fischer A, Thrasher AJ, Galy A, Cavazzana M. Outcomes following gene therapy in patients with severe Wiskott-Aldrich syndrome. JAMA. 2015 Apr 21;313(15):1550-63. doi: 10.1001/jama.2015.3253. PMID 25898053
- [Background] Howe SJ, Mansour MR, Schwarzwaelder K, Bartholomae C, Hubank M, Kempski H, Brugman MH, Pike-Overzet K, Chatters SJ, de Ridder D, Gilmour KC, Adams S, Thornhill SI, Parsley KL, Staal FJ, Gale RE, Linch DC, Bayford J, Brown L, Quaye M, Kinnon C, Ancliff P, Webb DK, Schmidt M, von Kalle C, Gaspar HB, Thrasher AJ. Insertional mutagenesis combined with acquired somatic mutations causes leukemogenesis following gene therapy of SCID-X1 patients. J Clin Invest. 2008 Sep;118(9):3143-50. doi: 10.1172/JCI35798. PMID 18688286
- [Background] Braun CJ, Boztug K, Paruzynski A, Witzel M, Schwarzer A, Rothe M, Modlich U, Beier R, Gohring G, Steinemann D, Fronza R, Ball CR, Haemmerle R, Naundorf S, Kuhlcke K, Rose M, Fraser C, Mathias L, Ferrari R, Abboud MR, Al-Herz W, Kondratenko I, Marodi L, Glimm H, Schlegelberger B, Schambach A, Albert MH, Schmidt M, von Kalle C, Klein C. Gene therapy for Wiskott-Aldrich syndrome--long-term efficacy and genotoxicity. Sci Transl Med. 2014 Mar 12;6(227):227ra33. doi: 10.1126/scitranslmed.3007280. PMID 24622513
- [Background] Burroughs LM, Nemecek ER, Torgerson TR, Storer BE, Talano JA, Domm J, Giller RH, Shimamura A, Delaney C, Skoda-Smith S, Thakar MS, Baker KS, Rawlings DJ, Englund JA, Flowers ME, Deeg HJ, Storb R, Woolfrey AE. Treosulfan-based conditioning and hematopoietic cell transplantation for nonmalignant diseases: a prospective multicenter trial. Biol Blood Marrow Transplant. 2014 Dec;20(12):1996-2003. doi: 10.1016/j.bbmt.2014.08.020. Epub 2014 Sep 6. PMID 25196857
- [Background] Danylesko I, Shimoni A, Nagler A. Treosulfan-based conditioning before hematopoietic SCT: more than a BU look-alike. Bone Marrow Transplant. 2012 Jan;47(1):5-14. doi: 10.1038/bmt.2011.88. Epub 2011 Apr 11. PMID 21478921
- [Background] Moshous D, Callebaut I, de Chasseval R, Corneo B, Cavazzana-Calvo M, Le Deist F, Tezcan I, Sanal O, Bertrand Y, Philippe N, Fischer A, de Villartay JP. Artemis, a novel DNA double-strand break repair/V(D)J recombination protein, is mutated in human severe combined immune deficiency. Cell. 2001 Apr 20;105(2):177-86. doi: 10.1016/s0092-8674(01)00309-9. PMID 11336668
- [Background] Rivera-Munoz P, Abramowski V, Jacquot S, Andre P, Charrier S, Lipson-Ruffert K, Fischer A, Galy A, Cavazzana M, de Villartay JP. Lymphopoiesis in transgenic mice over-expressing Artemis. Gene Ther. 2016 Feb;23(2):176-86. doi: 10.1038/gt.2015.95. Epub 2015 Oct 1. PMID 26361272
- [Background] Cavazzana M, Six E, Lagresle-Peyrou C, Andre-Schmutz I, Hacein-Bey-Abina S. Gene Therapy for X-Linked Severe Combined Immunodeficiency: Where Do We Stand? Hum Gene Ther. 2016 Feb;27(2):108-16. doi: 10.1089/hum.2015.137. PMID 26790362
- [Background] Long-Boyle JR, Savic R, Yan S, Bartelink I, Musick L, French D, Law J, Horn B, Cowan MJ, Dvorak CC. Population pharmacokinetics of busulfan in pediatric and young adult patients undergoing hematopoietic cell transplant: a model-based dosing algorithm for personalized therapy and implementation into routine clinical use. Ther Drug Monit. 2015 Apr;37(2):236-45. doi: 10.1097/FTD.0000000000000131. PMID 25162216
- [Background] Romero Z, Campo-Fernandez B, Wherley J, Kaufman ML, Urbinati F, Cooper AR, Hoban MD, Baldwin KM, Lumaquin D, Wang X, Senadheera S, Hollis RP, Kohn DB. The human ankyrin 1 promoter insulator sustains gene expression in a beta-globin lentiviral vector in hematopoietic stem cells. Mol Ther Methods Clin Dev. 2015 Apr 22;2:15012. doi: 10.1038/mtm.2015.12. eCollection 2015. PMID 26029723
- [Background] French D, Sujishi KK, Long-Boyle JR, Ritchie JC. Development and validation of a liquid chromatography-tandem mass spectrometry assay to quantify plasma busulfan. Ther Drug Monit. 2014 Apr;36(2):169-74. doi: 10.1097/01.ftd.0000443060.22620.cd. PMID 24625541
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Sherman SA, Burwinkle TM, Dickinson PE, Dixon P. The PedsQL Family Impact Module: preliminary reliability and validity. Health Qual Life Outcomes. 2004 Sep 27;2:55. doi: 10.1186/1477-7525-2-55. PMID 15450120
- [Background] Stoto MA. The accuracy of population projections. J Am Stat Assoc. 1983 Mar;78(381):13-20. doi: 10.1080/01621459.1983.10477916. PMID 12265583
- [Background] Casella G. Refining binomial confidence intervals. Canadian Journal of Statistics 14(2): 113-129, 1986.
- [Background] Mamcarz E, Zhou S, Lockey T, Abdelsamed H, Cross SJ, Kang G, Ma Z, Condori J, Dowdy J, Triplett B, Li C, Maron G, Aldave Becerra JC, Church JA, Dokmeci E, Love JT, da Matta Ain AC, van der Watt H, Tang X, Janssen W, Ryu BY, De Ravin SS, Weiss MJ, Youngblood B, Long-Boyle JR, Gottschalk S, Meagher MM, Malech HL, Puck JM, Cowan MJ, Sorrentino BP. Lentiviral Gene Therapy Combined with Low-Dose Busulfan in Infants with SCID-X1. N Engl J Med. 2019 Apr 18;380(16):1525-1534. doi: 10.1056/NEJMoa1815408. PMID 30995372
- [Background] Cowan MJ, Yu J, Facchino J, Fraser-Browne C, Sanford U, Kawahara M, Dara J, Long-Boyle J, Oh J, Chan W, Chag S, Broderick L, Chellapandian D, Decaluwe H, Golski C, Hu D, Kuo CY, Miller HK, Petrovic A, Currier R, Hilton JF, Punwani D, Dvorak CC, Malech HL, McIvor RS, Puck JM. Lentiviral Gene Therapy for Artemis-Deficient SCID. N Engl J Med. 2022 Dec 22;387(25):2344-2355. doi: 10.1056/NEJMoa2206575. PMID 36546626